CLINICAL TRIAL: NCT01718574
Title: Feasibility, Acceptability and Efficacy of Bibliotherapy for Patients With Cancer: a Randomized Control Trial
Brief Title: Bibliotherapy for Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Cedars CanSupport, Hope & Cope (Unknown)
Responsible Party: Principal Investigator, Dr. Annett Korner, PhD, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2888
Record Dates: First submitted 2012-10-24; First posted 2012-10-31 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Cancer
Keywords: self-help book; support service
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-help book (Experimental)
  Interventions: Other: Self-help book
- Usual Care Control (No Intervention)

INTERVENTIONS:
Other: Self-help book — Participants have 6 weeks to complete a 12 chapter self-help workbook. The workbook addresses: (i) The enhancement of a sense of personal control; and (ii) The learning of emotional and instrumental coping responses
  Arms: Self-help book

SUMMARY:
The purpose of this study is to examine the efficacy of a self-help workbook in enhancing a sense of empowerment, coping, quality of life and reducing distress for patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* been diagnosed with cancer
* can read English

Exclusion Criteria:

-participating in the "Think Smart, Live Well" group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
change in Health Education Impact Questionnaire scores | pre-intervention (week 0), post intervention (week 6), follow-up (week 10)

SECONDARY OUTCOMES:
change in Ways of Coping Questionnaire - Cancer Version & Hospital Anxiety and Depression Scale scores | pre-intervention (week 0), post intervention (week 6), follow-up (week 10)

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - MUHC Cedars CanSupport, Montreal, Quebec
  - Hope & Cope, JGH, Montreal, Quebec